CLINICAL TRIAL: NCT02233686
Title: A Double-blind, Randomised, Placebo-controlled, Crossover Study to Assess the Efficacy of XEN-D0501, a Transient Receptor Potential Vanilloid Receptor 1 (TRPV1) Antagonist, in Reducing the Frequency of Cough in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: A Study to Assess the Efficacy of XEN-D0501 in Reducing the Cough Frequency in Patients With COPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xention Ltd (Industry)
Collaborators: Ario Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XEN-D0501-CL-05
Record Dates: First submitted 2014-08-29; First posted 2014-09-08 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- XEN-D0501 (Experimental): 4mg BID Days 1-13, 4mg once daily (OD) Day 14
  Interventions: Drug: XEN-D0501
- Placebo to Match (Placebo Comparator): BID Days 1-13, once daily (OD) Day 14
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XEN-D0501
  Arms: XEN-D0501
Drug: Placebo
  Arms: Placebo to Match

SUMMARY:
The purpose of this study is to determine the effectiveness of XEN-D0501 over placebo in reducing the daytime cough frequency in patients with chronic obstructive pulmonary disease (COPD).

The effectiveness of XEN-D0501 placebo in reducing capsaicin cough responses, objective 24-hour cough frequency, hourly change in cough frequency, cough severity (via visual analogue scale [VAS]), urge to cough (via VAS), global rating of change scale, Clinical COPD Questionnaire (CCQ), Leicester Cough Questionnaire (LCQ), and St George's Respiratory Questionnaire (SGRQ-C) will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Male/female subjects aged 40 or over with COPD

Exclusion Criteria:

* Clinically significant medical history
* Abnormal laboratory results, ECGs or vital signs

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-02; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline at the end of each treatment period in objective daytime cough frequency | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Medicines Evaluation Unit, Manchester, United Kingdom